CLINICAL TRIAL: NCT04949165
Title: Iron Supplementation and Nutritional Counseling Interventions to Improve Availability and Safety of Blood in Ghana
Brief Title: Bloodsafe Ghana- Iron and Nutritional Counseling Strategy Pilot Study
Acronym: BLIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Blood Service Ghana (Other); University of Ghana Medical School (Other); Liverpool School of Tropical Medicine (Other); Syracuse University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 326045 - UG3HL151599; UG3HL151599 (NIH)
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Iron-deficiency Anemia; Iron-deficiency
Keywords: Blood donation
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron Supplementation (Experimental)
  Interventions: Dietary Supplement: Iron Supplementation
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Iron Supplementation — low dose ferrous sulphate (65mg elemental iron) supplements
  Arms: Iron Supplementation

SUMMARY:
This pilot study has 2 components: 1) a cross-sectional assessment designed to estimate the prevalence of anaemia leading to donor deferral, the prevalence of iron deficiency (ID) and iron deficiency anaemia (IDA) among first-time donors, and 2) a longitudinal 2-arm parallel groups trial among first- time voluntary donors that compares haemoglobin levels at 4 months among those with ID or IDA who receive iron supplementation to those without ID or IDA who do not receive iron supplementation. A structured questionnaire will be used to extract demographic characteristics. Participants will be followed for a total of 6 months with study visits at 2, 4 and 6 months after the baseline assessments. Blood draws for full blood count (FBC), peripheral film comment, malaria rapid diagnostic tests (RDT) and ferritin assessment will occur at baseline and all follow-up visits. In addition, we will use a qualitative approach to identify barriers and facilitators of blood donation and the use of dietary and iron supplementation strategies to address iron deficiency and/or anaemia. This will involve conducting focus group discussions during the last month of the intervention and key informant interviews.

Expected Outcomes The expected outcomes of the study have been grouped into two, primary and secondary. Primary Outcome will be haemoglobin level after 4 months. Secondary Outcomes are A. Change in haemoglobin levels B. Diagnosis of ID or IDA at 4 months C. Serum ferritin concentration after 4 months of intervention D. Acceptability of iron supplementation among participants and stakeholders E. Incidence of gastrointestinal adverse events F. Incidence of suspected malaria or bacterial infections G. Incidence of ID and IDA H. Successful return (non-deferred) to the blood donor pool after intervention within 6 months of enrolment I. Key barriers and facilitators of intervention implementation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged between 17 and 60 years who weigh at least 50kg.
* Pass pre-donation screening using the NBSG standardised donor screening questionnaire for medical conditions and lifestyle risks for transfusion transmissible infections
* Vital signs must meet the NBSG requirement for blood donation: systolic and diastolic blood pressures between 90-140 mmHg and 60- 90 mmHg, respectively; pulse rate between 50-100 bpm; non-contact forehead temperature not exceeding 37.5°C; meeting acceptable requirements for skin lesions, needle marks and physical appearance.
* Must be willing and able to give study consent or assent.
* Intend to remain in the study location/site during the entire length of the study.

Exclusion Criteria:

* Persons who have used iron supplementation within the past one month.
* Participant reports having previously donated blood.
* Evidence for a TTI at baseline among those who successfully donated.
* Evidence of Malaria and helminthic infections at baseline
* Participants who have Hb <10g/dl at screening

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 223 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ghana Medicial School, Department of Haematology, Accra, Ghana

IPD SHARING:
Plan to Share IPD: No
The BLOODSAFE project is committed to quickly sharing results and data. Papers will be submitted summarizing the primary results of the BLOODSAFE studies once the analysis is complete. These results will be published in major scientific journals and presented at scientific meetings.

REFERENCES:
- [Derived] Segbefia C, Telke S, Olayemi E, Ward C, Asamoah-Akuoko L, Appiah B, Yawson AE, Tancred T, Adu-Afarwuah S, Benneh-Akwasi Kuma A, Acquah ME, Ofori-Acquah SF, Adongo PB, Ametorwo R, Bates I, Reilly C, Dei-Adomakoh Y; BLOODSAFE Ghana Investigators. Deferrals for Low Haemoglobin and Anaemia Among First-Time Prospective Blood Donors in Southern Ghana: Results From the BLOODSAFE Ghana-Iron and Nutritional Counselling Strategy Pilot (BLIS) Study. Adv Hematol. 2025 May 6;2025:9971532. doi: 10.1155/ah/9971532. eCollection 2025. PMID 40365600

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Standard of care
Period: Overall Study
Arm/Group | Iron Supplementation | Control
Started | 105 | 118
Completed | 74 | 56
Not Completed | 31 | 62

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iron Supplementation | Control | Total
Number analyzed (Participants) | 105 | 118 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.70 (2.51) | 20.14 (3.09) | 19.93 (2.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 61 | 140
  Male | 26 | 57 | 83
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Akan | 55 | 57 | 112
  Ewe | 16 | 28 | 44
  Dagbani | 1 | 2 | 3
  Ga/Dangbe | 26 | 19 | 45
  Hausa | 0 | 2 | 2
  Other | 7 | 10 | 17
Current student [Count of Participants; unit: Participants]
  No | 3 | 2 | 5
  Yes | 102 | 116 | 218
National Blood Service Ghana deferral decision [Count of Participants; unit: Participants]
  Deferred | 40 | 3 | 43
  Not deferred | 65 | 115 | 180
Haemoglobin from FBC (g/dL) [Mean (Standard Deviation); unit: g/dL] | 11.25 (0.91) | 13.39 (1.26) | 12.38 (1.54)
Ferritin (log(ferritin + 1) [Mean (Standard Deviation); unit: ug/L] | 3.54 (0.87) | 4.21 (0.67) | 3.89 (0.84)
History of blood loss in the last 3 months [Count of Participants; unit: Participants] — Defined as donor reporting any of the following within the last 3 months: bleeding piles, stomach ulcer, bled from injury, surgery or treatment for malaria.
  Participants
    No | 78 | 78 | 156
    Yes | 27 | 40 | 67
Siblings with known related anaemia [Count of Participants; unit: Participants]
  No | 104 | 117 | 221
  Yes | 1 | 1 | 2
Heavy, frequent or long duration periods among menstrating women [Count of Participants; unit: Participants] — Defined as self-report of heavy periods, periods every 3 weeks or periods lasting longer than 10 days.
  Participants
    No | 40 | 37 | 77
    Yes | 37 | 25 | 62
    Not Applicable (Male or women who are no longer menstruating) | 28 | 56 | 84
Body mass index (kg/mˆ2) [Mean (Standard Deviation); unit: kg/mˆ2] | 24.12 (8.83) | 23.07 (3.31) | 23.57 (6.53)
Systolic blood pressure (mm Hg) [Mean (Standard Deviation); unit: mm Hg] | 116.35 (10.76) | 117.89 (11.08) | 117.17 (10.93)
Diastolic blood pressure (mm Hg) [Mean (Standard Deviation); unit: mm Hg] | 76.17 (7.94) | 76.92 (9.13) | 76.57 (8.58)
Number of meals yesterday [Count of Participants; unit: Participants]
  0 (fasting) | 1 | 0 | 1
  1 meal | 10 | 6 | 16
  2 meals | 40 | 47 | 87
  3 or more meals | 54 | 65 | 119

OUTCOME MEASURES:

1. Primary Outcome: Haemoglobin Level
Description: Haemoglobin level at 4 months from the enrollment visit.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Iron Supplementation | Control
Number analyzed (Participants) | 56 | 74
g/dL | 11.35 (1.27) | 12.28 (1.46)
Statistical Analysis 1: Comparison: Iron Supplementation vs Control; Test type: Non-Inferiority — The study employed a non-inferiority design with a non-inferiority margin of 1 g/dL for haemoglobin levels at 4 months, a 1-sided alpha level of 0.025, at least 85% power and under the assumption that the true difference in the means was 0.3 g/dL. The estimated sample size also allowed for up to 10% loss to follow- up or iron supplementation for those initially not requiring supplements, thus the sample size was 292; p = 0.025, t-test, 1 sided — Non-inferiority threshold of -1 g/dL for the lower bound of the 97.5% CI

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 26 weeks.
Arm/Group | Iron Supplementation | Control
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/118
Other Adverse Events (participants affected / at risk) | 0/105 | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT04949165/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT04949165/SAP_001.pdf